CLINICAL TRIAL: NCT03815994
Title: Effects of Physical Therapy With Neuromuscular Electrical Stimulation in Critically Ill Patients: a Randomised Crossover Clinical Trial Protocol.
Brief Title: Neuromuscular Electrical Stimulation in Critically Ill Patients.
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: This study had to be suspended due to COVID-19 Pandemic.
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ada Clarice Gastaldi, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: USP 2018-1
Record Dates: First submitted 2018-11-13; First posted 2019-01-25 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Critical Care; Rehabilitation
Keywords: Physical therapy modalities,; Electric stimulation therapy; Indirect calorimetry

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: group 1 (Experimental): Neuromuscular Electrical Stimulation (NMES) and after decubitus position with the limbs raised without NMES.
  Interventions: Device: Neuromuscular Electrical Stimulation
- group 2 (Sham Comparator): Decubitus Position with the limbs raised withou tNeuromuscular Electrical Stimulation and after Neuromuscular Electrical Stimulation.
  Interventions: Device: Neuromuscular Electrical Stimulation

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation — This device produces a muscle contraction in response to a externally generated low-voltage electric impulse, which is conducted through electrodes placed on the skin over the muscle group to be stimulated.
  Other Names: Functional Electrical Stimulation

SUMMARY:
The study will investigate the effects of neuromuscular electrical stimulation (NMES) in critically ill patients. The objective of this study will be investigate the effects of neuromuscular electrical stimulation (NMES) in critically ill patients.

DETAILED DESCRIPTION:
The study will investigate the effects of neuromuscular electrical stimulation (NMES) in critically ill patients. It will be a randomised crossover clinical trial. Thirty-one patients will enrolled. Patients will be selected, randomly, to the intervention Protocol (decubitus position with the limbs raised and NMES) and control (decubitus position with the limbs raised without NMES).The patients will be allocated in Group 1 (intervention and control) or group 2 (control and intervention) with a wash-out period of 4 to 6 hours between them.

The main outcome will be metabolic data. Linear mixed model will be used for analysis of dependent variables and estimated values of the mean of the differences of each effect.

The results of this study will allow better understanding of the metabolic effects of NMES in patients critically ill.

ELIGIBILITY:
Inclusion Criteria:

* All patients that will be admitted to the intensive care unit
* Hemodynamic stability
* Mechanical ventilation.

Exclusion Criteria:

1. In general:

   * a. Pregnant women
   * b. Brain death
   * c. Neuromuscular diseases
   * d. Use of pre-existing neuromuscular blocker in the last 24 hours, prior to the study protocol.
2. Contraindications for the use of NMES:

   * a. Fractures
   * b. Burns
   * c. Skin lesions
   * d. Systemic vascular impairment diseases such as systemic lupus erythematosus, thromboembolic disease, deep vein thrombosis (which was not therapeutically anticoagulated for a time greater than 36 hours)
   * e. Lower limb amputations
   * f. Cardiac pacemaker,
   * g. Thrombocytopenia less than 20,000/mm3
   * h. BMI greater than 35 kg/m2
   * i. Important lower extremity oedema
   * j. Agitation and/or signs of pain during the electrical stimulation.
3. Contraindications to begin or continue NMES procedure:

   * a. Mean arterial blood pressure less than 65 mmHg
   * b. Use of vasopressor >50% of themaximum dose (dopamine >12.5 μg/kg per minute; vasopressin >0.02U/min and norepinephrine >1 μg/kg per minute),
   * c. Heart rate <50 or >140bpm
   * d. Arrhythmias with hemodynamic consequences
   * e. Myocardial ischemia,
   * f. Temperature <34 or >39oC
   * g. Intracranial pressure >20 cmH2O
   * h. Decrease in 10% of SpO2 baseline value or <88% for more than one minute.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2018-11-13 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2021-01-29 (Estimated)

PRIMARY OUTCOMES:
Change of Oxygen consumption (VO2),from baseline and interventions. | VO2 will be taken during the each intervention, it will be taken only the first day
  Change of Oxygen consumption (VO2) will be evaluated by calorimetry

SECONDARY OUTCOMES:
Change of Carbon dioxide production (VCO2) from baseline and interventions. | VCO2 will be taken during the each intervention, it will be taken only the first day
  Change of Carbon dioxide production (VCO2) will be evaluated by calorimetry

OTHER OUTCOMES:
Change of Resting energy expenditure (REE) from baseline and interventions. | REE will be taken during the each intervention, it will be taken only the first day
  Change of Resting energy expenditure (REE) will be evaluated by calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Ada C Gastaldi, PhD, Principal Investigator — Ribeirao Preto Medicine School-University of São Paulo
Locations (1):
- Clinics Hospital, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, will be available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available immediately following publication and for five years.
Access Criteria: The data will be available from the principal investigator upon reasonable request.

REFERENCES:
- [Derived] Lago AF, Basile-Filho A, de Oliveira AS, de Souza HCD, Dos Santos DO, Gastaldi AC. Effects of physical therapy with neuromuscular electrical stimulation in acute and late septic shock patients: A randomised crossover clinical trial. PLoS One. 2022 Feb 17;17(2):e0264068. doi: 10.1371/journal.pone.0264068. eCollection 2022. PMID 35176099